CLINICAL TRIAL: NCT02962830
Title: Assessment of Fetal and Maternal Sufentanil Pharmacokinetics After Intra-amniotic Injection
Brief Title: Sufentanil Pharmacokinetics After Intra Amniotic Injection
Acronym: 2IAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014_19; 2015-001721-16 (EudraCT Number)
Record Dates: First submitted 2016-08-17; First posted 2016-11-11 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Prenatal Diagnosis
Keywords: fetal pain; fetal analgesia
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sufentanil (Experimental)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — intra-amniotic injection of 10 micrograms of Sufentanil

SUMMARY:
The fetus may be exposed during pregnancy to nociceptive stimuli because of fetal pathology (e.g., malformation) or a diagnostic or therapeutic procedure.

To date, there is very little data and no consensus on fetal analgesia. The aim of the investigators study is to evaluate the pharmacokinetics of Sufentanil after intra amniotic injection.

ELIGIBILITY:
Inclusion Criteria:

* Termination of pregnancy for fetal malformation
* Gestational age > 24 weeks of gestation

Exclusion Criteria:

* Multiple pregnancy
* Allergy or contraindication to sufentanil
* Morphinic addiction
* fetal gastroschisis, omphalocele or swallowing disorder
* maternal cardiac or respiratory distress

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
fetal plasma concentrations | at 30 minutes after intra-amniotic injection
  fetal plasma concentrations of morphine derivatives by Ultrahigh Pressure Liquid Chromatography (UPLC) with mass spectometry (Triple Quadrupole Detector)

SECONDARY OUTCOMES:
Maternal plasma concentrations | at 30 minutes and at 1, 2, 4, 8, 24 hours after intra-amniotic injection
  Maternal plasma concentrations of morphine derivatives by Ultrahigh Pressure Liquid Chromatography (UPLC) with mass spectometry (Triple Quadrupole Detector)
amniotic fluid concentrations | Immediately within 5 min after intra-amniotic injection
  The amniotic fluid concentrations of morphine derivatives by Ultrahigh Pressure Liquid Chromatography (UPLC) with mass spectometry (Triple Quadrupole Detector)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique HOUFFLIN-DEBARGE, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No